CLINICAL TRIAL: NCT06187753
Title: Sensory Processing Issues in Children With Eosinophilic Esophagitis
Brief Title: Sensory Processing Issues in Eosinophilic Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Assistant Professor, Gazi University
Other Study IDs: 100714
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Eosinophilic Esophagitis; Sensory Disorder
MeSH Terms: conditions — Eosinophilic Esophagitis; Sensation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Eosinophilic Esophagitis: Children with Eosinophilic Esophagitis The first group will consist 30 children with definite EoE diagnoses who were between ages 3 and 10 years. The Sensory Profile will used to evaluate sensory processing. This questionnaire will be completed by parents who record a child's responses to sensory events in daily life.
  Interventions: Diagnostic Test: Sensory Profile
- Children with Typically Developing: Typically Developing Children The second group will consist of 30 children with typically developing who were between ages 3 and 10 years. The Sensory Profile will used to evaluate sensory processing. This questionnaire will be completed by parents who record a child's responses to sensory events in daily life.
  Interventions: Diagnostic Test: Sensory Profile

INTERVENTIONS:
Diagnostic Test: Sensory Profile — The Sensory Profile has 125 items that represent 14 functions of sensory processing and allows parents to report on their child's behavior.

SUMMARY:
Feeding dysfunction and/or dysphagia are the main symptoms of eosinophilic esophagitis (EoE). Also, these symptoms may be a part of sensory processing disorders. Therefore, the present study compared sensory processing abilities between children with EoE and typically developing (TD) controls.

DETAILED DESCRIPTION:
Eosinophilic Esophagitis (EoE) is a chronic allergic/immune condition of the esophagus that affects all ages, from infancy through adulthood. The chronic inflammation can lead to symptoms that vary with age. It is critically important to know symptoms in the infancy/toddler period because in this period, they can't express symptoms directly. The frequent symptoms seen in this period are; vomiting, refusing sucking and eating, failure to thrive, and abdominal pain. School-aged children with EoE have decreased appetite, recurrent abdominal pain, vomiting, food impaction, and dysphagia. Feeding dysfunction (feeding refusal, slowly eating, picky eater, etc..) is one of the trouble issues in this period. Children who can't experience different texture (especially solid) and tastes of foods keep on eating with their same safe feeding habits. Whereas experiences gained in early childhood period form the basis of sensory and motor development. As currently known, humans have eight senses (visual, auditory, gustatory, olfactory, tactile, proprioception, vestibular, and interoception). Each sense is unique, a form of information and nourishment for the nervous system. In the meantime, it is crucial to receive, interpret, and integrate all this information from all these senses at a time. Sensory integration (SI) is the term used for the brain processing information that comes through the senses. The SI begins in the womb as the fetal brain senses the movements. Childhood activities and play lead to a lot of sensory integration as the child organizes the sensations of his body and gravity, along with sight and sound. If there is a problem in any sense, such as receiving or interpreting, the SI process can be interrupted, and this may result in sensory processing disorder (SPD). It is crucial to notice SPD in childhood because SPD can affect a child's development and education (learning, reading, math, visual and auditory perception, and skilled motor tasks).

Food intake is one of the most multi-sensory daily experiences (sight, smell, taste, sounds, texture of food) for both children and adults. In children with EoE, feeding dysfunction (vomiting, food impaction, regurgitation..) can affect the oral sensory system. Even considering that all the senses work in interaction, more senses can be affected.

To date, there is no study that has investigated sensory processing issues in children with EoE. Therefore, the present study aimed to compare sensory processing between children with EoE and healthy controls and also examine the correlations between sensory processing and disease characteristics among children with EoE.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of EoE
* being between 3 and 10 years

Exclusion Criteria:

* having acute illnesses
* having any other chronic diseases

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with eosinophilic esophagitis and age-matched typically developing peers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile | Baseline
  The questionnaire has 125 items that represent 14 functions of sensory processing and allows parents to report on their child's behavior. The questionnaire uses a five-point rating scale, with a score of '1' indicating always or 100%, '2' indicating frequently or at least 75%, '3' indicating occasionally or 50%, '4' indicating seldom or 25%, and '5' indicating never or 0%. Six categories defined by the Sensory Profile are related to sensory processing areas, while five categories relate to sensory modulation, and the last three categories reflect social-emotional responses related to sensory processing. The test also provides nine sensory profile factor scores that reflect sensory processing styles.

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation Recruiting Ankara, Turkey, 06500, Ankara, Turkey (Türkiye)